CLINICAL TRIAL: NCT04707209
Title: Intravitreal Injection of Sirolimus in the Treatment of Aggressive Retinal Astrocytic Hamartoma
Brief Title: Sirolimus for Retinal Astrocytic Hamartoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Ashwin Mallipatna, Paediatric Ophthalmologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000072947
Record Dates: First submitted 2020-12-16; First posted 2021-01-13 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Retinal Astrocytic Hamartoma
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravitreal Sirolimus (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — An intravitreal injection of 20 µL of drug will be given through the pars plana of the eye. The injected eye will be treated with topical antibiotic and steroid eye drops prescribed for 7 to 10 days after the injection. The first injection will only be provided into the worse eye despite both eyes showing signs of exudation. Injection into the other eye will be considered only two months after the safety of this first injection is determined.
  Safety and efficacy of treatment will be determined by repeat eye examinations in the eye clinic one day, one week and one month after each injection.
  The interval between injections is roughly suggested to be between 3 to 8 weeks based on the drug deposit present in the eye. A total of 3-12 injections will be given per eye, over 6-24 months.
  Other Names: DE-109

SUMMARY:
A single patient study using intravitreal Sirolimus to treat a patient with multiple retinal astrocytic hamartomas (RAH) of both eyes.

DETAILED DESCRIPTION:
Retinal astrocytic hamartomas (RAH) are benign tumors of glial cells arising from astrocytes in the nerve-fiber layer of the retina. They are often associated with tuberous sclerosis complex (TSC) and, more rarely, neurofibromatosis type 1 (NF1). RAH may be caused by dysregulated tumor suppressors genes TSC1 or TSC2, which play a role in cell cycle regulation in retinal astrocytes via the PDGF-signalling pathway. Downregulation of TSC1 or TSC2 can result in hyperactivation of mTOR. Sirolimus is an inhibitor of mTOR, therefore inhibiting cell growth and proliferation of astrocytes. Systemic mTOR inhibitors (sirolimus and everolimus) have shown impressive reduction in the size of RAH in animal models and many human case series.

This single patient study is investigating the use of concurrent oral and intravitreal Sirolimus to treat a patient with multiple retinal astrocytic hamartomas (RAH) of both eyes to improve intraocular response and reduce duration of treatment. The patient has no other clinical features suggestive of neurofibromatosis and a presumed diagnosis of tuberous sclerosis is being considered, with only two hypopigmented skin lesions noted.

ELIGIBILITY:
Single case diagnosed with multiple retinal astrocytic hamartomas (RAH) of both eyes with imminent threat to vision.

Ages: 15 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Size of Retinal Astrocytic Hamartomas compared to baseline | 21 months
  Measured by ophthalmic imaging
Amount of retinal exudate compared to baseline | 21 months
  Measured by ophthalmic imaging
Retinal detachment progression/regression compared to baseline | 21 months
  Measured by ophthalmic imaging

SECONDARY OUTCOMES:
Visual acuity compared to baseline | 21 months
  Measured using logMAR virtual activity test

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No